CLINICAL TRIAL: NCT02569970
Title: Efficacy of Fluoxetine Against Seizure-induced Central Apneas : a Randomized Placebo-controled Double-blind Trial.
Brief Title: Efficacy of Fluoxetine Against Seizure-induced Central Apneas
Acronym: FLUOXETINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-562
Record Dates: First submitted 2015-09-24; First posted 2015-10-07 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Epilepsy; Ictal/Post-ictal Hypoxemia
Keywords: Epilepsy; SUDEP; fluoxetine; placebo; SpO2
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLUOXETINE (Active Comparator): 4 weeks of treatment before video-EEG monitoring
  Interventions: Drug: fluoxetine 20 mg
- PLACEBO (Placebo Comparator): 1 month of treatment before EEG video.
  Interventions: Drug: placebo 20 mg

INTERVENTIONS:
Drug: fluoxetine 20 mg — Fluoxetine 20 mg per day during 4 weeks prior to video-EEG, then continued during video-EEG.
  At the end of video-EEG, and according to patient's decision, treatment was either progressively withdrawn (1 week at 10 mg per day and then 1 week at 5 mg per day), or replaced by fluoxetine 20 mg open-label.
  Arms: FLUOXETINE
Drug: placebo 20 mg — Placebo 20 mg per day during 4 weeks prior to video-EEG, then continued during video-EEG.
  At the end of video-EEG, and according to patient's decision, treatment was either progressively withdrawn (1 week at 10 mg per day and then 1 week at 5 mg per day), or replaced by fluoxetine 20 mg open-label.
  Arms: PLACEBO

SUMMARY:
Sudden unexpected death in epilepsy (SUDEP) is a tragic outcome of seizure disorders that primarily affect young adults suffering from refractory epilepsy. In this population, SUDEP incidence is estimated at 0.5%. While the mechanisms of SUDEP are not completely understood, it appears that the majority of such death occurs in the immediate aftermath of a general tonic-clonic seizure.

There is currently no validated preventive treatment for SUDEP. Some evidence suggest that modulation of the serotoninergic tone, and more specifically selective serotonin recapture inhibitor (SSRI) such as fluoxetine, might prevent SUDEP. Indeed, fluoxetine prevents seizure-induced lethal central apneas in DBA/2 and DBA/1 mice, one of the few animal models of SUDEP. Furthermore, serotoninergic bulbar nuclei are known to play a major role in the control of breathing, especially during sleep and in response to repeated hypoxia.

In patients with epilepsy undergoing in-hospital video-EEG monitoring, about one third of seizures are associated with decrease in SpO2 <90%, an abnormality suspected to represent a risk factor of SUDEP. In a retrospective uncontrolled study, patients treated with SSRIs displayed less frequent ictal/post-ictal hypoxemia than patients not taking SSRIs.

The investigators project aimed at testing whether fluoxetine can reduce the risk of ictal/post-ictal hypoxemia by performing a double-blind, randomized, placebo-controlled trial in patients undergoing video-EEG monitoring as part of the pre-surgical evaluation of their focal drug-resistant epilepsy.

ELIGIBILITY:
Inclusion Criteria:

Patient suffering from drug-resistant focal epilepsy

* Age ≥ 18 years
* Patient for whom a video-EEG monitoring of their seizures was scheduled as part of a pre-surgical assessment
* For women of childbearing age, a method of contraception considered effective by the investigator
* Patient who have given their written informed consent
* Patient accepting an interview with a psychologist and to be refered to a psychiatrist in the event that mood disorders were detected on mood scores and considered severe by the investigator and / or psychologist, leading to require psychiatric care or immediate antidepressant treatment
* Patient with a social security number

Exclusion Criteria:

* Age < 18 years

  * Patient under legal protection
  * Pregnant or breastfeeding women
  * Hypersensitivity to fluoxetine or its excipients
  * History of other serious side effects related to an earlier prescription of fluoxetine;
  * Current suicidal ideation or history of suicide attempt
  * Manic episode
  * Disruption of liver enzymes considered material by the investigator using the following criteria:

transaminases (ALT and AST)> 2N alkaline phosphatase (ALP)> 2N gamma glutamyl transpeptidase (GGT)> 5N (performed as part of routine monitoring of epileptic patients on antiepileptic treatment. Patients often exhibit changed deemed clinically insignificant due to the enzyme-inducing effect of these drugs)

* Renal failure with creatinine clearance <30 ml / min
* Acute heart disease
* Antidepressant treatment
* Other prohibited treatment (see detailed list in protocol).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Ictal/post-ictal hypoxemia | Duration of video-EEG following 4 weeks of fluoxetine treatment
  Percentage of patients with at least one seizure associated with ictal/post-ictal SpO2 <90% in the group treated with fluoxetine compared to that receiving placebo.

SECONDARY OUTCOMES:
Change in mood score with BDI-II score | After four weeks of treatment as compared to baseline
  Changes in score of BDI-II after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo
Change in mood score with NDDIE score | After four weeks of treatment as compared to baseline
  Changes in score of NDDIE after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo
Change in seizure frequency | After four weeks of treatment as compared to baseline
  Changes in seizure frequency after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo
Change in sleep disorders score with SASDQ score | After four weeks of treatment as compared to baseline
  Changes in score of SASDQ after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo
Change in sleep disorders score with EPWORTH score | After four weeks of treatment as compared to baseline
  Changes in score of EPWORTH after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo
Change in score of quality of life | After four weeks of treatment as compared to baseline
  Change in score of QOLIE-89 after four weeks of treatment as compared to baseline in the group treated with fluoxetine compared to that receiving placebo

CONTACTS AND LOCATIONS:
Overall Officials: Philippe RYVLIN, Professor, Study Director — Hospices Civils de Lyon
Locations (1):
- Service de Neurologie Fonctionnelle et d'Epileptologie, Hôpital Neurologique, Lyon, France